CLINICAL TRIAL: NCT02650193
Title: A Phase 1-2 Ascending Dose Study To Assess The Pharmacodynamics, Pharmacokinetics, And Safety Of Hsp-130 In Subjects With Non-metastatic Breast Cancer Following Single-dose And Multiple-dose Administration By Subcutaneous Injection
Brief Title: A Study Of The Safety And Effects Of One Or More Doses Of HSP-130 Injected Under The Skin In Women With Breast Cancer That Has Not Spread To Distant Sites In The Body.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZIN-130-1504; C1221002 (Other: Alias Study Number); 2015-002057-35 (EudraCT Number)
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Non-metastatic Breast Cancer
Keywords: HSP-130 Phase 1-2 Study in patients with Breast cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HSP-130 (Experimental): Cycle 0:
  Regimen A: HSP 130, 3 mg, single SC injection in the deltoid region (n = 6) Regimen B: HSP 130, 6 mg, single SC injection in the deltoid region (n = 6)
  Cycles 1-4:
  Regimen B (n = 12): HSP 130, 6 mg, single SC injection in the deltoid region, at least 24 hours after administration of chemotherapy in Cycle 1, Cycle 2, Cycle 3, and Cycle 4.
  Potential Regimen A (n = 12): 3 mg with background chemotherapy: Inclusion of this cohort will be based on assessment of comparability between Regimens A and B in Cycle 0 for ANC and CD34+ as defined above. If performed, this regimen will be HSP 130, 3 mg, single SC injection in the deltoid region, at least 24 hours after administration of chemotherapy in Cycle 1, Cycle 2, Cycle 3, and Cycle 4, as appropriate.
  Conditional Regimen C (12 mg):This cohort will not be initiated until data from cycle 0 for 3 mg and 6 mg and Cycles 1-4 for 6 mg has been reviewed and analyzed.
  Interventions: Drug: HSP-130

INTERVENTIONS:
Drug: HSP-130 — Dosage will vary per each cohort: (Five independent cohorts) Cycle 0 Regimen A - 3 mg Cycle 0 Regimen B - 6 mg Cycles 1-4 Regimen B - 6 mg Cycles 1-4 Regimen A (Potential)- 3 mg Cycles 1-4 Regimen C (Conditional)- 12 mg
  Other Names: Pegylated filgrastim

SUMMARY:
This is a study of how one or more injections of HSP-130 under the skin effect the white blood cell counts and drug levels in women with breast cancer that has not spread to distant sites in the body (non-metastatic). This will be studied in women before breast surgery or while receiving chemotherapy. Safety will also be studied.

Additionally, the purpose of this study is to evaluate the effects and safety of single and multiple doses of HSP-130 in subjects with non-metastatic breast cancer. This study will determine the dose to move forward for future clinical trials.

DETAILED DESCRIPTION:
This is an open-label, sequential enrollment study characterizing the pharmacodynamic (PD), pharmacokinetic (PK) and safety of HSP-130 in subjects with non-metastatic breast cancer who have not previously received chemotherapy at any point prior to enrollment in this study (ZIN-130-1504).

The purpose of this study is to evaluate the effects and safety of single and multiple doses of HSP-130 in subjects with non-metastatic breast cancer. This study will determine the dose to move forward for future clinical trials.

There are two aspects of the study. In the initial part of the study, 6 subjects will be sequentially enrolled to receive HSP-130 treatment (3 mg , or 6 mg by subcutaneous injection) during the period between biopsy and definitive surgery. This will determine whether 3 mg and 6 mg have similar or different effects on the PD variables (absolute neutrophil counts and CD34+ cell counts). This part of the study is referred to as Cycle 0 since study subjects will receive no chemotherapy while receiving HSP-130 until the effect of HSP-130 on the PD variables is known. A total of 12 subjects may be enrolled in Cycle 0.

The objective of Cycle 1-4 is to determine the dose to be taken forward to Phase 3 clinical trials. Cycles 1-4 subjects will receive HSP-130 after their definitive breast surgery at the time they receive TAC chemotherapy (docetaxel, doxorubicin, and cyclophosphamide). Subjects will receive up to 4 cycles of every 3 week TAC chemotherapy with HSP-130 given on Day 2 of the chemotherapy regimen.

* If the 3 mg dose is found to be inferior (potentially subtherapeutic) to the 6 mg dose in Cycle 0, only the 6 mg dose will be studied in Cycles 1-4 (n=12), when subjects receive concomitant chemotherapy.
* If the 3 mg dose is found to be comparable to the PD results obtained in Cycle 0 with 6 mg, the 3 mg dose (n=12) will also be studied in women receiving TAC chemotherapy.

Data from the HSP-130 6 mg regimen (plus 3 mg, as appropriate) will be analysed, discussed with the FDA and determination if a dose greater than 6 mg is appropriate to study (e.g., 12 mg). If all three doses are studied, a total enrollment of up to 36 subjects is projected for Cycles 1-4.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for study participation if all of the following criteria are met at Screening:

  1. Is informed, has been given ample time and opportunity to read about participation in the study and has signed and dated the written informed consent form approved by an Independent Ethics committee (IEC) prior to any study related activities
  2. Females ≥ 18 years
  3. Histologically confirmed and documented invasive breast cancer
  4. Breast cancer without evidence of distant metastases (Stage 4) based on staging work-up
  5. Chemotherapy naive, who have not received chemotherapy in the neoadjuvant setting and who are candidates for chemotherapy in the adjuvant setting of taxane/cyclophosphamide-based regimen, e.g., TAC, as background chemotherapy
  6. Zubrod/WHO/ECOG performance status ≤ 2
  7. Adequate bone marrow, hepatic, and renal function reserve as evidenced by:

     1. Hemoglobin ≥ 10 mg/dl
     2. ANC ≥ 1.5 x 10^9/L
     3. Platelet count of ≥ 100 x 10^9/L
     4. Total bilirubin ≤ 2 mg/dl
     5. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 3 x the upper limit of normal (ULN) of the reference lab
     6. Serum creatinine of ≤ 1.5 x ULN for reference lab or estimated glomerular filtration rate (eGFR) of ≥ 60 mg/min
  8. Body mass index (BMI) of 19 to 40 kg/m^2 , inclusive
  9. Subjects of childbearing potential, and their partners, agree to pregnancy prevention throughout the duration of the study (through the Follow-up Visit). Specific type of pregnancy prevention should be discussed with, and acceptable to, the treating oncologist in the context of the tumoral hormone receptor status. Subjects and their partners must agree to use of an effective method of contraception, to avoid impregnation of females throughout the course of the study

     Medically acceptable forms of birth control can include, with approval of the treating physician:
     1. Barrier methods (condom or diaphragm with spermicide)
     2. Intrauterine device (IUD)
     3. Hormone contraceptives (such as oral [pill], injection, skin patch, implant, cervical ring)
     4. Subjects using oral contraceptives must be on a stable regimen for at least 3 months prior to Screening. Sexually active subjects must use contraception while on HSP-130 from admission to the final Follow-up Visit
  10. Able to understand verbal or written instructions and comply with all study requirements, to communicate effectively with study personnel and is available for the planned duration of the study

Exclusion Criteria:

* A subject will NOT be eligible for study participation if any of the following criteria are met at Screening:

  1. Previous G-CSF exposure, including filgrastim, lenograstim, pegfilgrastim, lipegfilgrastim, granulocyte/macrophage colony stimulating growth factor (GM-CSF), or any other branded or biosimilar G-CSF
  2. Prior autologous stem cell harvest of any type
  3. Drug sensitivity, allergic reaction, or known hypersensitivity or idiosyncratic reaction to E. coli - derived proteins, filgrastim, other G-CSFs, or pegylated agents
  4. Known hypersensitivity to docetaxel, polysorbate 80, or doxorubicin
  5. For subjects receiving doxorubicin, no concurrent use of inhibitors and inducers of CYP3A4, CYP2D6, and/or P-gp or with trastuzumab due to increased risk of cardiac dysfunction
  6. Chemotherapy other than that included in this study (taxane/cyclophosphamide-based regimen, e.g., TAC or TC) or neoadjuvant chemotherapy; or known immunosuppressive agents including chronic oral corticosteroid use, or radiation therapy within 4 weeks of first dose of HSP-130, prior bone marrow or stem cell transplantation, or malignancy within 5 years
  7. Known HER2 + ( overexpressing breast cancer)
  8. Known triple negative (estrogen receptor-negative, progesterone receptor-negative and HER2-negative) breast cancer
  9. ≥ Grade 2 underlying neuropathy
  10. Current diagnosis of active tuberculosis or other severe infection, such as sepsis, abscesses or opportunistic infections
  11. Treatment with systemically active antibiotics within 72 hours before chemotherapy
  12. Known infection with HIV
  13. Known sickle cell disease
  14. Known severe persistent drug-induced myelosuppression
  15. New York Heart Association (NYHA) class III or IV heart failure, severe uncontrolled cardiac disease (unstable angina, clinically significant ECG abnormalities) or MI within the previous 6 months before the first administration of HSP-130
  16. Any malignancy other than breast cancer, with exception of adequately treated squamous or basal cell carcinoma of the skin or cervical carcinoma in situ, within 5 years before the first administration of the HSP-130
  17. Current or recent treatment (within 30 days before the first administration of the HSP-130) with any other investigational medicinal product
  18. Pregnancy or lactation; Subjects planning to be pregnant or to breastfeed before, during, or within 12 months after administration of the HSP-130 are not permitted to enroll in the study
  19. Received a live, live-attenuated, or non-live vaccine within 4 weeks before the first administration of the HSP-130
  20. Patient has evidence of any other coexisting disease or medical or psychological condition, metabolic dysfunction, physical examination finding or clinical lab finding giving reasonable suspicion of a disease or condition that contraindicated the use of an HSP-130, or patient is high risk for treatment complication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Hungary (3):
  - CRU Hungary Kft.,CRU Early Phase Unit, Miskolci Semmelweis Kórház és Egyetemi Oktató Kórház, Miskolc, BAZ Megye
  - Debreceni Egyetem Klinikai Központ, ÁOK, Onkológiai Klinika, Debrecen, Hajdú-bihar Megye
  - Országos Onkológiai Intézet, Budapest
- Spain (4):
  - Hospital Universitario Arnau de Vilanova, Lleida, Catalonia
  - Hospital Universitario de Fuenlabrada, Servicio de oncologia, Fuenlanbrada, Madrid
  - START Madrid - CIOCC, Unidad de fases 1 planta 3, Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Arnau de Vilanova. planta 6, unidad de Oncología, Valencia

REFERENCES:
- [Derived] Yao HM, Jones SR, Morales S, Moosavi S, Zhang J, Freyman A, Ottery FD. Phase I/II study to assess the clinical pharmacology and safety of single ascending and multiple subcutaneous doses of PF-06881894 in women with non-distantly metastatic breast cancer. Cancer Chemother Pharmacol. 2021 Dec;88(6):1033-1048. doi: 10.1007/s00280-021-04355-6. Epub 2021 Oct 7. PMID 34618197

RESULTS

PARTICIPANT FLOW:
Groups:
- Cycle 0: HSP-130 3mg: Participants who had not received background chemotherapy treatment in the study were administered a single dose of 3 milligram (mg) of HSP-130 subcutaneously (SC) at Day 1 of Cycle 0. Participants were followed approximately 30 days after last dose of study treatment.
- Cycles 0: HSP-130 6mg: Participants who had not received background chemotherapy treatment in the study were administered a single dose of 6 mg of HSP-130 SC at Day 1 of Cycle 0. Participants were followed approximately 30 days after last dose of study treatment.
- Cycles 1-4: HSP-130 6mg: Participants in Cycles 1-4 received background chemotherapy treatment at Day 1 and were administered a single dose of 6 mg of HSP-130 SC at Day 2 of Cycles 1-4 (each cycle was approximately 3 weeks if there were no chemotherapy treatment delays). Participants were followed approximately 30 days after last dose of study treatment.
Period: Overall Study
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Started | 6 | 6 | 13
Completed | 6 | 6 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study medication.
Groups:
- Cycle 0: HSP-130 3mg: Participants who had not received background chemotherapy treatment in the study were administered a single dose of 3 mg of HSP-130 SC at Day 1 of Cycle 0. Participants were followed approximately 30 days after last dose of study treatment.
- Total: Total of all reporting groups
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg | Total
Number analyzed (Participants) | 6 | 6 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (8.89) | 60.8 (13.60) | 55.1 (8.95) | 59.3 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 13 | 25
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 10 | 21
  Unknown or Not Reported | 0 | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 6 | 13 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Effect Curve for Absolute Neutrophil Count (AUECANC): Cycle 0
Description: Absolute neutrophil count (ANC) is a measure of the number of neutrophil granulocytes (also known as polymorphonuclear cells, PMN's, polys, granulocytes, segmented neutrophils or segs) present in the blood.
Time Frame: Cycle 0: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. This outcome measure was not planned to be analyzed for Cycles 1-4: HSP-130 6mg arm.
Measure: Mean (Standard Deviation); unit: hour*10^9 Neutrophils per Liter
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
hour*10^9 Neutrophils per Liter | 3900.482 (683.6870) | 5880.985 (1287.2887)

2. Primary Outcome: Area Under the Serum Concentration Time Curve From Time of Dose Administration to Time Infinity (AUCinf): Cycle 0
Description: AUCinf = Area under the serum concentration of HSP-130 versus time curve (AUC) from the time of dose administration to extrapolated infinite time (0-inf).
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: hour*picogram per milliliter (h*pg/mL)
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
hour*picogram per milliliter (h*pg/mL) | 1425862.2 (949518.8) | 5689476.1 (3757035.5)

3. Primary Outcome: Maximum Observed Serum Concentration (Cmax): Cycle 0
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
picogram per milliliter (pg/mL) | 38026.7 (28821.7) | 155766.7 (99051.8)

4. Primary Outcome: Duration of Severe Neutropenia (DSN): Cycle 1
Description: Severe Neutropenia was defined as grade 4 neutropenia in which the ANC was < 0.5 x10^9 per liter. DSN was defined as the days with grade 4 neutropenia (ANC < 0.5 x10^9/L).
Time Frame: Cycle 1: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. This outcome measure was not planned to be analyzed for Cycle 0: HSP-130 3mg and Cycle 0: HSP-130 6mg arms. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for the specified outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 12
days | 0.667 (0.9847)

5. Primary Outcome: Area Under the Serum Concentration Time Curve From Time of Dose Administration to Time of Last Measurable Concentration (AUCt): Cycle 1 and Cycle 4
Description: AUC0-t= Area under the serum concentration of HSP-130 versus time curve from the time of dose administration to time of last quantifiable concentration (0-t).
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
h*pg/mL
  Cycle 1 | 10084193.7 (14047222.7)
  Cycle 4 | 6017621.6 (5920395.4)

6. Primary Outcome: Maximum Observed Serum Concentration (Cmax): Cycle 1 and Cycle 4
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
pg/mL
  Cycle 1 | 118130.8 (119028.6)
  Cycle 4 | 95200.0 (93544.1)

7. Secondary Outcome: Maximum Effect for Absolute Neutrophil Count (ANC_Emax): Cycle 0
Description: ANC was a measure of the number of neutrophil granulocytes (also known as polymorphonuclear cells, PMN's, polys, granulocytes, segmented neutrophils or segs) present in the blood.
Time Frame: Cycle 0: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: *10^9 Neutrophils per Liter
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
*10^9 Neutrophils per Liter | 24.512 (6.0710) | 43.257 (5.5683)

8. Secondary Outcome: Time of Maximum Effect for Absolute Neutrophil Count (ANC_Tmax): Cycle 0
Description: as for outcome 7
Time Frame: Cycle 0: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
hour | 71.950 [48.00 to 144.10] | 47.800 [46.90 to 48.30]

9. Secondary Outcome: Area Under the Effect Curve for CD34+ (AUECCD34+): Cycle 0
Time Frame: Cycle 0: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*cells per microliter (h*cells/ mcL)
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
hour*cells per microliter (h*cells/ mcL) | 1749.523 (1022.3037) | 2752.198 (2152.8794)

10. Secondary Outcome: Maximum Effect for CD34+ Count (CD34+_Emax): Cycle 0
Time Frame: Cycle 0: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/mcL)
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
cells per microliter (cells/mcL) | 13.970 (6.8536) | 27.343 (18.4805)

11. Secondary Outcome: Time of Maximum Effect for CD34+ Count (CD34+ Tmax): Cycle 0
Time Frame: Cycle 0: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
hour | 96.000 [48.00 to 96.10] | 96.600 [95.80 to 191.30]

12. Secondary Outcome: Area Under the Effect Curve for Absolute Neutrophil Count From Time of Dose Administration to Time Infinity (AUEC_ANC Inf): Cycle 0
Description: ANC is a measure of the number of neutrophil granulocytes (also known as polymorphonuclear cells, PMN's, polys, granulocytes, segmented neutrophils or segs) present in the blood.
Time Frame: Cycle 0: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for the specified outcome measure.
Measure: Mean (Standard Deviation); unit: hour*10^9 Neutrophils per Liter
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 5 | 6
hour*10^9 Neutrophils per Liter | 5254.288 (1699.7088) | 6576.165 (1821.9919)

13. Secondary Outcome: Area Under the Effect Curve From Time of Dose Administration to Time Infinity for CD34 + (AUEC_CD34+ Inf): Cycle 0
Time Frame: Cycle 0: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. This outcome measure was not planned to be analyzed for Cycles 1-4: HSP-130 6mg arm. Here "Overall number of participants analyzed" signifies number of participants evaluable for the specified outcome measure.
Measure: Mean (Standard Deviation); unit: hour*cells per microliter (h*cells/mcL)
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 5
hour*cells per microliter (h*cells/mcL) | 1835.221 (1036.6473) | 3159.470 (2197.4774)

14. Secondary Outcome: Area Under the Serum Concentration Time Curve From the Time of Dose Administration to the Time of Last Measurable Concentration (AUCt): Cycle 0
Description: as for outcome 5
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
h*pg/mL | 1410202.6 (948443.5) | 5677700.3 (3756049.2)

15. Secondary Outcome: Time To Achieve Maximum Serum Concentration (Tmax): Cycle 0
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: hour
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
hour | 12.0 [12 to 12] | 23.5 [6 to 24]

16. Secondary Outcome: Elimination Half-Life (t1/2): Cycle 0
Description: t1/2 is the time taken for plasma concentration of HSP 130 to reduce by 50 percent (%) of its initial value.
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
hour | 50.0 (15.5) | 48.8 (12.5)

17. Secondary Outcome: Elimination Rate Constant (λz): Cycle 0
Description: Elimination rate constant was defined as the rate at which the drug was removed from the body.
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
per hour | 0.015 (0.0051) | 0.015 (0.0041)

18. Secondary Outcome: Apparent Clearance (CL/F): Cycle 0
Description: Clearance of a drug was defined as the rate at which a drug was metabolized or eliminated by normal biological processes.
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: milliliter per hour (mL/h)
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
milliliter per hour (mL/h) | 4235.6 (4714.4) | 1655.9 (1242.6)

19. Secondary Outcome: Protein-Content Corrected Area Under the Serum Concentration Time Curve From Time of Dose Administration to Time Infinity (AUCinf): Cycle 0
Description: The protein-content correction was conducted for AUCinf parameter: Protein-content corrected AUCinf = Nominal Protein-content AUCinf / (Actual protein concentration/10.0 mg/mL).
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
h*pg/mL | 1440264.8 (959109.9) | 5689476.1 (3757035.5)

20. Secondary Outcome: Protein-Content Corrected Area Under the Serum Concentration Time Curve From Time of Dose Administration to Time of Last Measurable Concentration (AUCt): Cycle 0
Description: The protein-content correction was conducted for AUCt parameter: Protein-content corrected AUCt= Nominal Protein-content AUCt / (Actual protein concentration/10.0 mg/mL).
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
h*pg/mL | 1424447.1 (958023.7) | 5677700.3 (3756049.2)

21. Secondary Outcome: Protein-Content Corrected Maximum Observed Serum Concentration (Cmax): Cycle 0
Description: The protein-content correction was conducted for Cmax parameter: Protein-content corrected Cmax = Nominal Protein-content Cmax / (Actual protein concentration/10.0 mg/mL).
Time Frame: Cycle 0: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg
Number analyzed (Participants) | 6 | 6
pg/mL | 38410.8 (29112.8) | 155766.7 (99051.8)

22. Secondary Outcome: Duration of Severe Neutropenia (DSN): Cycle 4
Description: Severe Neutropenia was defined as grade 4 neutropenia in which the ANC was < 0.5 x10^9/L. DSN was defined as the days with grade 4 neutropenia (ANC < 0.5 x10^9/L).
Time Frame: Cycle 4: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. This outcome measure was not planned to be analyzed for Cycle 0: HSP-130 3mg and Cycle 0: HSP-130 6mg arms. Here, 'Overall number of participants analyzed" signifies number of participants evaluable for the specified outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 12
days | 0.667 (0.9847)

23. Secondary Outcome: Absolute Neutrophil Count Nadir Concentration: Cycle 1 and Cycle 4
Description: Nadir was defined as the lowest count for ANC concentration reported after first dose of study treatment.
Time Frame: Cycle 1 and 4: Predose (0 hour), 48, 96, 144, 192, 240, and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. This outcome measure was not planned to be analyzed for Cycle 0: HSP-130 3mg and Cycle 0: HSP-130 6mg arms.
Measure: Mean (Standard Deviation); unit: *10^9 Neutrophils per Liter
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
*10^9 Neutrophils per Liter
  Cycle 1 | 1.132 (1.1480)
  Cycle 4 | 1.623 (1.8364)

24. Secondary Outcome: Time of ANC Nadir Concentration: Cycle 1 and Cycle 4
Description: Time of ANC Nadir (in hours) was defined as the time from the first dose of study treatment on Day 2 of Cycle 1 and 4 to the time the lowest value was recorded.
Time Frame: Cycle 1 and 4: Predose (0 hour), 48, 96, 144, 192, 240, and 312 hours post-dose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
hour
  Cycle 1 | 129.231 (23.0585)
  Cycle 4 | 142.154 (65.3323)

25. Secondary Outcome: Area Under the Effect Curve (AUEC_ANCt): Cycle 1 and Cycle 4
Description: as for outcome 12
Time Frame: Cycle 1 and 4: Predose (0 hour), 48, 96, 144, 192, 240, and 312 hours post-dose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hour*10^9 Neutrophils per Liter
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
hour*10^9 Neutrophils per Liter
  Cycle 1 | 2540.285 (854.2237)
  Cycle 4 | 3186.542 (1362.0079)

26. Secondary Outcome: Area Under the Effect Curve for Absolute Neutrophil Count From Time of Dose Administration to Time Infinity (AUEC_ANC Inf): Cycle 1 and Cycle 4
Description: as for outcome 1
Time Frame: Cycle 1 and 4: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. Here, "number analyzed" field signifies that the number of participants were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: hour*10^9 Neutrophils per Liter
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
hour*10^9 Neutrophils per Liter
  Cycle 1: number analyzed (Participants) | 8
  Cycle 1 | 5636.963 (1974.1635)
  Cycle 4: number analyzed (Participants) | 7
  Cycle 4 | 12399.370 (18345.3366)

27. Secondary Outcome: Incidence of Febrile Neutropenia: Cycle 1 and Cycle 4
Description: Febrile Neutropenia was defined as tympanic or axillary body temperature greater than (>) 38.5 °C for >1 hour and ANC less than (<) 1.0 *10^9/L.
Time Frame: Cycle 1 and 4: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
participants
  Cycle 1 | 1
  Cycle 4 | 0

28. Secondary Outcome: Incidence of Severe Neutropenia: Cycle 1 and Cycle 4
Description: Severe Neutropenia was defined as grade 4 neutropenia in which the ANC was < 0.5 x10^9/L.
Time Frame: Cycle 1 and 4: Predose (0 hour), 48, 96, 144, 192, 240, and 312 hours post-dose
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
participants
  Cycle 1 | 5
  Cycle 4 | 5

29. Secondary Outcome: Time to ANC Recovery: Cycle 1 and Cycle 4
Description: Time to ANC recovery was defined as the time from documentation of the first day with ANC greater than equal to (>=) 2.0 x10^9/L after any day with ANC <2.0 x10^9/L.
Time Frame: Cycle 1 and 4: Predose (0 hour), 48, 96, 144, 192, 240 and 312 hours post-dose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
days
  Cycle 1 | 2.615 (1.7097)
  Cycle 4 | 2.000 (1.633)

30. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time of Dose Administration to Time Infinity (AUCinf): Cycle 1 and Cycle 4
Description: AUC0-inf = Area under the serum concentration versus time curve (AUC) from the time of dose administration to extrapolated infinite time (0-inf).
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. Here, 'number analyzed' field signifies that the number of participants were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
h*pg/mL
  Cycle 1 | 10093213.5 (14047936.2)
  Cycle 4: number analyzed (Participants) | 12
  Cycle 4 | 6425013.3 (6000938.3)

31. Secondary Outcome: Time To Achieve Maximum Serum Concentration (Tmax): Cycle 1 and Cycle 4
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: hour
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
hour
  Cycle 1 | 24.1 [12 to 48]
  Cycle 4 | 23.5 [6 to 142]

32. Secondary Outcome: Elimination Half-Life (t1/2): Cycle 1 and Cycle 4
Description: t1/2 is the time taken for plasma concentration of a drug to reduce by 50% of its initial value.
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. Here 'number analyzed' signifies number of participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
hour
  Cycle 1 | 30.7 (10.8)
  Cycle 4: number analyzed (Participants) | 12
  Cycle 4 | 29.5 (9.5)

33. Secondary Outcome: Elimination Rate Constant (λz): Cycle 1 and Cycle 4
Description: Elimination rate constant was defined as the rate at which the drug was removed from the body.
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. Here, 'number analyzed' signifies number of participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
per hour
  Cycle 1 | 0.026 (0.0099)
  Cycle 4: number analyzed (Participants) | 12
  Cycle 4 | 0.025 (0.0060)

34. Secondary Outcome: Apparent Clearance (CL/F): Cycle 1 and Cycle 4
Description: CL/F was defined as a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
mL/h
  Cycle 1 | 1326.8 (1010.2)
  Cycle 4: number analyzed (Participants) | 12
  Cycle 4 | 2342.8 (2043.8)

35. Secondary Outcome: Protein-Content Corrected Area Under the Serum Concentration Time Curve From Time of Dose Administration to Time of Last Measurable Concentration (AUCt): Cycle 1 and Cycle 4
Description: as for outcome 20
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
h*pg/mL
  Cycle 1 | 10087666.8 (14045724.4)
  Cycle 4 | 6045733.4 (5955438.5)

36. Secondary Outcome: Protein-Content Corrected Area Under the Serum Concentration Time Curve From Time of Dose Administration to Time Infinity (AUCinf): Cycle 1 and Cycle 4
Description: as for outcome 19
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication. Here 'number analyzed' signifies number of participants evaluable at the specified timepoints only.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
h*pg/mL
  Cycle 1 | 10096698.3 (14046434.6)
  Cycle 4: number analyzed (Participants) | 12
  Cycle 4 | 6454443.8 (6037499.6)

37. Secondary Outcome: Protein-Content Corrected Maximum Observed Serum Concentration (Cmax): Cycle 1 and Cycle 4
Description: as for outcome 21
Time Frame: Cycle 1 and 4: Predose (0 hour), 6, 12, 24, 48, 96, 144, 192, 240 and 312 hours post-dose
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 13
pg/mL
  Cycle 1 | 118173.0 (119004.2)
  Cycle 4 | 95670.1 (94209.4)

38. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in participants who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment Emergent Adverse Event (TEAE) was adverse event that started or worsened in severity after the HSP-130 administration up to and including 30 days post HSP-130 administration (up to Day 94). AEs included both serious and non-serious.
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
Participants
  AEs | 6 | 6 | 13
  SAEs | 0 | 0 | 2

39. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) of Special Interest
Description: AEs of Special Interest (AESI) included Potential Allergic Reactions, Splenomegaly, Splenic Rupture, Acute Respiratory Distress Syndrome, Alveolar Hemorrhage, Hemoptysis, Leukocytosis, Thrombocytopenia, Capillary Leak Syndrome, Cytokine Release Syndrome, Cutaneous Vasculitis and Glomerulonephritis.
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
Participants | 0 | 2 | 2

40. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria: hematology (hemoglobin, hematocrit, platelet count, white blood cell count, neutrophils); chemistry (alkaline phosphatase, glucose, lactate dehydrogenase, alanine aminotransferase, aspartate aminotransferase, albumin, creatinine and gamma-glutamyl transpeptidase, blood urea nitrogen, total protein, phosphate, and uric acid); urinalysis. The clinical laboratory results and patterns observed were consistent with the known therapeutic response and the safety profile for the US and EU approved pegylated filgrastim (Neulasta).
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
Participants | 6 | 6 | 13

41. Other Pre Specified Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Vital sign assessment included body temperature (tympanic or axillary), heart rate (sitting), blood pressure (sitting systolic and diastolic), and respiratory rate. Clinically significant abnormality was based upon investigator's discretion.
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
Participants | 0 | 0 | 0

42. Other Pre Specified Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities
Description: Physical examination included physical assessment of the spleen. Clinically significant abnormality was based on investigator's discretion.
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
Participants | 0 | 0 | 0

43. Other Pre Specified Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Clinically significant abnormality was based upon investigator's discretion.
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
Participants | 0 | 0 | 0

44. Other Pre Specified Outcome: Number of Participants With At Least 1 Concomitant Medication
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
Participants | 6 | 6 | 13

45. Other Pre Specified Outcome: Duration of Exposure to Study Drug Medication
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: days
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
days | 3.00 [3.00 to 3.00] | 6.00 [6.00 to 6.00] | 24.0 [24.0 to 24.0]

46. Other Pre Specified Outcome: Number of Participants With Positive Anti-pegfilgrastim (Anti-drug) Antibodies
Time Frame: Baseline up to approximately Day 94
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cycle 0: HSP-130 3mg | Cycles 0: HSP-130 6mg | Cycles 1-4: HSP-130 6mg
Number analyzed (Participants) | 6 | 6 | 13
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to approximately Day 94
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Groups:
- Cycle 0: HSP-130 6mg: Participants who had not received background chemotherapy treatment in the study were administered a single dose of 6 mg of HSP-130 SC at Day 1 of Cycle 0. Participants were followed approximately 30 days after last dose of study treatment.
- Cycle 1-4: HSP-130 6mg: Participants in Cycles 1-4 received background chemotherapy treatment at Day 1 and were administered a single dose of 6 mg of HSP-130 SC at Day 2 of Cycles 1-4 (each cycle was approximately 3 weeks if there were no chemotherapy treatment delays). Participants were followed approximately 30 days after last dose of study treatment.
Arm/Group | Cycle 0: HSP-130 3mg | Cycle 0: HSP-130 6mg | Cycle 1-4: HSP-130 6mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/13
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 0: HSP-130 3mg (N=6) | Cycle 0: HSP-130 6mg (N=6) | Cycle 1-4: HSP-130 6mg (N=13)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 0: HSP-130 3mg (N=6) | Cycle 0: HSP-130 6mg (N=6) | Cycle 1-4: HSP-130 6mg (N=13)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 4
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 7
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 2
Chest discomfort (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 3
Inflammation (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arachnoid cyst (Nervous system disorders) | 1 | 0 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 4 | 5
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 8
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT02650193/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT02650193/SAP_001.pdf